CLINICAL TRIAL: NCT00888641
Title: A Pilot Study of Renal Hypothermia During Partial Nephrectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Bradley Leibovich, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-007979
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Kidney Neoplasm
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normothermia (No Intervention): After arterial clamping, no ice slush will be used
- Hypothermia (Experimental): After arterial clamping, the kidney will be surrounded in ice slush for 10 minutes
  Interventions: Procedure: Hypothermia

INTERVENTIONS:
Procedure: Hypothermia — Surround kidney in ice slush for 10 minutes after arterial clamping
  Arms: Hypothermia

SUMMARY:
Renal hypothermia may preserve renal function in patients who require partial nephrectomy. In preparation for a definitive randomized controlled trial this pilot study will assess feasibility and variance data to be used for sample size estimation

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with a renal mass deemed amenable to an open partial nephrectomy regardless of stage or histology.
2. Bilateral renal function on radiographic imaging.
3. Willing to consent to randomization.
4. Willing to comply with study protocol.

Exclusion Criteria:

1. Anatomically or functionally solitary kidney
2. Multiple renal tumours
3. Bilateral renal tumours
4. Life expectancy < 3 months as deemed by treating physician
5. Age less than 18 years old
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
measures of renal function uCrCl be performed for estimation of renal function | 3 months

SECONDARY OUTCOMES:
Post-operative complication | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States